CLINICAL TRIAL: NCT05632094
Title: The Efficacy of L-Carnitine in the Management of Acute Clozapine Intoxication
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, zahraa khalifa sobh, Assistant Professor of Forensic Medicine and Clinical Toxicology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2302
Record Dates: First submitted 2022-11-10; First posted 2022-11-30 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Clozapine Poisoning
Keywords: Clozapine Toxicity; Clozapine Poisoning; Clozapine Intoxication; L-Carnitine; Antioxidant; Egypt
MeSH Terms: interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: Clinical controlled randomized clinical trial (phase II) will be conducted in Poison Center. The total required sample size is 40 patients who suffer from acute clozapine intoxication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Group (No Intervention): This group will comprise 20 patients who will receive conventional supportive care for the treatment of acute clozapine toxicity that include the following:
  * Airway: maintaining clear patent airways.
  * Breathing: oxygen inhalation, respiratory support whenever required (mechanical ventilation).
  * Circulation: intravenous fluids, and symptomatic treatment according to ECG abnormalities.
  * Decontamination: administration of activated charcoal (1 gm/kg).
- L-Carnitine Group (Experimental): This group will comprise 20 patients who will receive conventional supportive care (same as group 1), in addition to IV L-carnitine
  Interventions: Dietary Supplement: L-Carnitine

INTERVENTIONS:
Dietary Supplement: L-Carnitine — The clozapine-intoxicated patients will receive conventional supportive care in addition to IV L-carnitine with a loading dose of 100 mg/kg IV over 30-60 min (maximum 6 g) and the maintenance dose was 50 mg/kg IV every 8 h.
  Arms: L-Carnitine Group

SUMMARY:
Clozapine is a dibenzodiazepine that is used atypical antipsychotic drug. Clozapine-induced cytotoxicity could be attributed to increases in reactive oxygen species (ROS) that oxidize mitochondrial proteins and disrupt cellular respiration.

L-Carnitine (4-N-trimethylammonium-3-hydroxybutyric acid) is an endogenous mitochondrial membrane compound that is essential for the normal functions of mitochondria. L-Carnitine is an effective ROS scavenger that prevents lipid peroxidation.

In an animal study, it was observed that clozapine decrease L-Carnitine level in plasma which results in metabolic disorders. Subsequently, the use of supplementation L-Carnitine was recommended to attenuate clozapine-induced side effects.

An in-vitro study investigated the cytotoxic effects of clozapine on human lymphocytes and the possible protective role of L-Carnitine, the results revealed that clozapine-induced cytotoxicity attributed to oxidative stress and mitochondrial dysfunction which significantly improved upon L-Carnitine administration.

In clinical toxicology, acute clozapine toxicity results in significant morbidities and mortalities in absence of a specific antidote. Therefore, it is essential to adopt pharmaceutical intervention based on the proposed mechanism of clozapine-induced cytotoxicity.

The objective of the current research is to assess the potential beneficial effects of L-Carnitine on the acute clozapine poisoning outcome.

The study will include patients with moderate and severe acute clozapine poisoning. The patient's condition will be assessed on admission using a Poisoning Severity Score.

Patients with acute clozapine poisoning will be assigned randomly into two groups; the Conventional group and the L-Carnitine group. Then, all patients will be closely followed up for vital signs, Glasgow Coma Scale, and Electrocardiogram. Clinical and laboratory reassessments will be performed. Lastly, the outcomes will be assessed and statistical analysis of the results will be performed.

Ethical approval was obtained from the Research Ethics Committee of the Faculty of Medicine, Alexandria University. This Ethics Committee is constituted and operates according to ICH GCP Guidelines and applicable local and institutional regulations and guidelines that govern the Ethics Committees operation. Written informed consent will be obtained from clozapine-intoxicated patients or their guardians (minors or those with disturbed mental status). Full details regarding the study's aim and procedures will be provided to all participants. A code number will be assigned to ensure confidentiality and anonymous analysis of data.

DETAILED DESCRIPTION:
Study design:

Clinical controlled randomized clinical trial (phase II) will be conducted in Poison Center. The total required sample size is 40 patients, similar to the sample size calculated in the clinical trial that verified the efficacy of IV lipid emulsion in managing clozapine toxicity.

The diagnosis will be based on the history of intake of a large dose of clozapine along with the presence of the pill container. The diagnosis of acute clozapine toxicity will be supported by the clinical findings that include significant central nervous system depression, hypotension, tachycardia, and prolongation of QT interval.

All patients will be subject to the following:

* History taking: Sociodemographic data, the amount of ingested drug, time past since ingestion, pre-hospital management, current medical complaints, past medical and surgical history.
* Clinical assessment: Glasgow coma scale, vital signs, and general examination).
* Laboratory investigations that included: arterial blood gases (ABG), complete blood count, serum sodium and potassium levels, blood glucose level, liver functions (bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT)), renal functions (urea, creatinine, blood urea nitrogen (BUN)) and cardiac enzymes.
* Electrocardiogram.
* Calculation of Poisoning Severity Score (PSS) that classifies poisoning severity as none (0), minor (1), moderate (2), severe (3), and fatal (4).

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with moderate and severe acute clozapine poisoning. The patient's condition will be assessed on admission using a Poisoning Severity Score.

Exclusion criteria:

* When the diagnosis of acute clozapine poisoning is unconfirmed.
* Patients with significant comorbidities, especially advanced neurological and cardiac diseases.
* Patients that ingest other drugs other than clozapine.
* Patients who presented late to the poison center (>24 hr) following clozapine intake.
* Patients received treatment before hospital admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | up to 14 days
  Death
Neurotoxicity | up to 14 days
  Changes in Scores of Glasgow Coma Scale (GCS). GCS is scored between 3 and 15, with 3 being the worst and 15 the best.
Cardiotoxicity | up to 14 days
  Changes in the rate of sinus rhythm and QT interval in Electrocardiogram

SECONDARY OUTCOMES:
Intensive care unit admission | up to 14 days
  Number of patients who need intensive care unit admission
Duration of hospital stay | up to 14 days
  Hours passed since admission till discharge or death

IPD SHARING:
Plan to Share IPD: Undecided
The confidentiality of the personal data of participants will be maintained. I intended to publish the current study in an international academic journal. Then, the published data could be accessed and used for any purpose.

REFERENCES:
- [Background] Abbas MF, Abbas AH. Clozapine-induced myocarditis in rats: role of L-carnitine in protection. The Egypt J. Forensic Sci. Appli. Toxicol. 2016; 16(1): 141-157. doi: 10.21608/ejfsat.2016.39958
- [Background] Wang W, Bai M, Jiang T, Li C, Li P, Zhou H, Wang Z, Li L, Jiang H. Clozapine-induced reduction of l-carnitine reabsorption via inhibition/down-regulation of renal carnitine/organic cation transporter 2 contributes to liver lipid metabolic disorder in mice. Toxicol Appl Pharmacol. 2019 Jan 15;363:47-56. doi: 10.1016/j.taap.2018.11.007. Epub 2018 Nov 19. PMID 30465787
- [Background] Pourahmad J, Salimi A, Imani F, Jamali Z, Ahvar N. The clozapine-induced toxicity via induction of oxidative stress and mitochondrial dysfunction in human blood lymphocytes and protecting role of L-Carnitine. Int. pharm. acta. 2020;3(1), 3e9:1-9. https://doi.org/10.22037/ipa.v3i1.32179
- [Background] Sherif NA, El-Banna AS, ElBourini MM, Khalil NO. Efficacy of L-carnitine and propranolol in the management of acute theophylline toxicity. Toxicol Res (Camb). 2020 Mar 11;9(1):45-54. doi: 10.1093/toxres/tfaa002. eCollection 2020 Feb. PMID 32440337
- [Background] Elgazzar FM, Elgohary MS, Basiouny SM, Lashin HI. Intravenous lipid emulsion as an adjuvant therapy of acute clozapine poisoning. Hum Exp Toxicol. 2021 Jul;40(7):1053-1063. doi: 10.1177/0960327120983873. Epub 2021 Jan 5. PMID 33401984